CLINICAL TRIAL: NCT03678701
Title: Effects of Protein Supplementation on Fat Mass Loss in Free Living Individuals With Overweight and Obesity - A Randomized Controlled Trial
Brief Title: Protein Supplementation and Fat Mass Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Emily Dhurandhar, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2018-126
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: whey protein; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein group (Experimental): The protein group will consume 30g of 100% whey protein shake 1 hour before lunch and before dinner, for 12 weeks
  Interventions: Dietary Supplement: Pre-meal 100% whey protein intake
- Control group (No Intervention): Control group will not consume any protein supplements. They will continue the usual feeding habits

INTERVENTIONS:
Dietary Supplement: Pre-meal 100% whey protein intake — Participants in the protein group will be provided 100% whey protein powder and will be advised to drink 30g of protein dissolved in 237ml (8oz) of water, one hour before lunch and dinner.
  Arms: Protein group

SUMMARY:
Investigators examined the associations between whey protein supplementation before meals with energy balance and body composition.

DETAILED DESCRIPTION:
Increase intake of dietary protein has been shown to have a role in weight loss and weight management since it affects satiety, thermogenesis, energy efficiency, and body composition. However, the effects of long-term protein supplementation on body fat mass in free living individuals with overweight and obesity are not known. This knowledge is important because people are more likely to take a protein supplement and expect to achieve fat loss without any other life style modification. Our research question is, whether consumption of whey protein supplements prior to main meals will reduce body weight and body fat without other intentional behavioral changes. We hypothesize that, addition of a 30g protein drink (100% whey isolate) 1 hour before lunch and dinner would promote negative energy balance, leading to body fat reduction in free living individuals with overweight and obesity in the absence of any other lifestyle changes. Our specific aims are: (1) To determine the impact of long-term protein supplementation on energy expenditure and body composition; (2) To determine the impact of long-term protein supplementation in free living condition on satiety and hunger; and (3) To determine the impact of long-term protein supplementation on physical activity and muscle strength. To test our hypothesis, we will conduct a 12-week, two parallel group randomized controlled trial with an additional baseline week. The intervention group will be advised to consume 30g whey protein shake 1 hour before lunch and before dinner for 12 weeks while the control group will not consume protein shakes. Both groups will continue usual dietary habits and physical activity. We will measure food intake using 3-day dietary records pre-intervention, and during intervention at week 7, and 12. Physical activity will be monitored using a hip worn accelerometer pre-intervention and during 6th week of intervention. Measurements taken pre-intervention, at the end of 6th week and at the end of 12th week include body weight, body composition using dual energy x-ray absorptiometry and bioelectrical impedance analysis. Resting metabolic rate will be measured using indirect calorimetry pre- and post-intervention. Between-meal satiety and hunger will be measured using 100 mm Visual Analog Scales at 6am, 11am, I hour after lunch, 6pm, 1 hour after dinner at baseline, day 14th, 43th and 83rd.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19-55 years
* Body mass index more than or equal to 23 kg/m2 for Asians and more than or equal to 25 kg/m2 for other ethnic groups up to 40 kg/m2
* Individuals who are able to speak, read and write in English

Exclusion Criteria:

* Lactose intolerance
* Food allergies to milk products
* Religious affiliations that include specific food guidelines.
* Participation in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months or planning to enroll in those within next 3 months
* History of prior surgical procedure for weight control or planning to have one within next 3 months
* Weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss.
* Current smoker or quit smoking less than 6 months prior.
* Any major disease, including:

  * Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
  * Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
  * Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months.
  * Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
  * Active renal disease.
  * Lung disease: chronic obstructive airway disease requiring use of oxygen.
  * Diagnosed diabetes (type 1 or 2).
  * On medication that may not be absorbed while on whey protein supplements: Levodopa, alendronate and Albendazole
  * Diagnosed hypertension or resting blood pressure more than 140/90
  * Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.
  * Zung Self-Rating Depression Scale score is >42 and Eating Attitudes Test score to ensure that our participants do not have symptoms of depression
  * History of or current eating disorders, or an Eating Attitudes Test (EAT-26) score >20
  * Conditions or behaviors likely to affect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; another household member is a participant or staff member in the trial; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating clinics before trial completed; unable to walk 0.25 mile in 10 minutes.
  * Currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months.
  * A recent or ongoing problem with drug abuse or addiction.
  * Excessive alcohol intake, either acute or chronic, defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months; or 3) other evidence available to clinic staff.
  * Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.
* Currently taking medication that suppresses or stimulates appetite or that affects body weight, including oral anti-diabetic medications.
* Anyone currently taking statins
* Pregnancy and childbearing: currently pregnant or less than 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the course of the trial; unwilling to take adequate contraceptive measures if potentially fertile.
* Not willing to stop taking protein supplements for the next 3 months, if selected for the control
* Engaged in aerobic physical activity (brisk walking, jogging, and running) for more than 30 minutes per day for 5 times per week or performing any resistance training
* Ratings for the supplement taste is 5 or more on a Likert Scale from 1= "Dislike extremely" to 9= "Like extremely" after tasting the protein shake
* Any other conditions which in opinion of the investigators that would adversely affect the conduct of the trial will also be excluded

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Group differences in change in body fat mass | Baseline, end of 6th week and end of 12th week of intervention period
  Fat mass will be measured using a Lunar Dual X-Ray Absorptiometry Scanner (GE Medical Systems) and the Imp SFB7 BIS (ImpediMed Ltd, Australia) at baseline, and at end of the treatment period. The outcome to be compared between groups will be change in percent fat mass from baseline to post treatment.

SECONDARY OUTCOMES:
Group differences in change in physical activity energy expenditure | Baseline and week 7 of the intervention period
  Participants will be instructed to wear a tri-axial accelerometer (AntiGraph GT3X+, Pensacola, FL) on their right hip during waking hours for 7 days. Accelerations will be summed over 1 minute epochs and 60 minutes will be used to determine non-wear time. Using the Freedson VM3 Combination algorithm (42) in Actilife v6.13.3, accelerometer data will be processed to yield estimates of daily and weekly PAEE for each treatment period. Participants will be asked to wear an accelerometer and keep a log of their daily activities that include planned exercise for seven days during week 3 of the protocol.
Group differences in changes in meal satiety and hunger | Baseline, day 14, 43 and 83 of intervention period
  Satiety and hunger will be measured using 100 mm Visual Analog Scales anchored by "not at all" to "extremely" in response to questions about hunger, fullness, desire to eat, and ability to eat more just before consuming before and after meals. Participants will be asked to fill out these questionnaires at 6am, 11am, I hour after lunch, 6pm, 1 hour after dinner.
Group differences in change in resting Metabolic Rate | Baseline, and at end 12 weeks of intervention period
  Resting metabolic rate will be measured by indirect calorimetry using the Cosmed's FitMateTM (COSMED, Italy) metabolic system using a canopy dilution set-up.
Group differences in changes in food intake | Baseline, at week 7, and at week 12 of intervention period
  Food intake will be studied over 3 days (one weekend and 2 weekdays) Dietary data will be used to calculate energy intake and macronutrient distribution of participant diets using the USDA nutrient database.
Group differences in changes in grip strength | Baseline and after the 6th and 12th week of intervention.
  Grip strength will be measured using the Lafayette Hand Grip Dynamometer
Group differences in change in lean mass | Baseline and after 6th and 12th week of intervention
  Lean mass will be measured using a Lunar Dual X-Ray Absorptiometry Scanner

CONTACTS AND LOCATIONS:
Overall Officials: Emily J (806)834-6556, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No